CLINICAL TRIAL: NCT06419439
Title: Ketamine-assisted Integrative Treatment for Veterans With Chronic Low Back Pain and Comorbid Depression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: NURP-001-23F; IK2CX002646-01A2 (NIH)
Record Dates: First submitted 2024-04-23; First posted 2024-05-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low Back Pain; Depression
Keywords: Feasibility Studies; Pilot Projects; Randomized Controlled Trials; Clinical trials; Psychosocial Intervention; Narrative Medicine; Narrative Therapy; Ketamine; Ketamine, therapeutic use; Veterans; Veterans, Research Subjects; Low Back Pain, Recurrent/Chronic; Depression; Hallucinogens, Therapeutic Use
MeSH Terms: conditions — Depression; Narrative Medicine; Low Back Pain; Recurrence; Bronchiolitis Obliterans Syndrome | interventions — Ketamine; Exercise; Methods

STUDY DESIGN:
Intervention Model Description: This study will occur in two phases which will occur sequentially and have different designs. The initial phase is a single-arm open-label, nonrandomized, non-blinded pilot study (n=5). The objective is to develop and assess initial feasibility of study procedures and obtain participant feedback through semi-structured exit interviews. The subsequent phase, informed by these findings, will consist of a single-blind, two-arm, pilot feasibility randomized controlled trial (RCT) (n=44, 22 per arm) which will (a) assess feasibility benchmarks and (b) collect outcome data that will be used to calculate sample size to power a larger RCT.
Who Masked: Participant
Masking Description: Participants in the second phase only will be blinded to the arm (intervention+minimally enhanced usual care vs minimally enhanced usual care alone).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Open label, single arm pilot (Other): Initial phase: A small open-label, single arm pilot study (n=5) will be conducted to develop and assess initial feasibility of study procedures and obtain participant feedback through semi-structured exit interviews. All participants in this open-label single arm pilot will receive the intervention (ketamine infusions followed by the brief behavioral intervention). There will be no control condition, randomization, or blinding.
  Interventions: Drug: Ketamine hydrochloride; Behavioral: Brief narrative intervention
- Intervention + Minimally Enhanced Usual Care (Experimental): Second phase: Intervention arm of a single-blind, two-arm, pilot feasibility randomized controlled trial (RCT) (n=44, 22 per arm) which will (a) assess feasibility benchmarks and (b) collect outcome data that will be used to calculate sample size to power a larger RCT.
  Minimally Enhanced Usual Care will consist of educational reading materials regarding chronic back pain and depression.
  Interventions: Drug: Ketamine hydrochloride; Behavioral: Minimally Enhanced Usual Care; Behavioral: Brief narrative intervention
- Minimally Enhanced Usual Care Only (Active Comparator): Second phase: Control arm of a single-blind, two-arm, pilot feasibility randomized controlled trial (RCT) (n=44, 22 per arm) which will (a) assess feasibility benchmarks and (b) collect outcome data that will be used to calculate sample size to power a larger RCT.
  Minimally Enhanced Usual Care will consist of educational reading materials regarding chronic back pain and depression.
  Interventions: Drug: Ketamine hydrochloride; Behavioral: Minimally Enhanced Usual Care

INTERVENTIONS:
Drug: Ketamine hydrochloride — Participants in Arms 1, 2, and 3 will receive four twice-weekly ketamine hydrochloride intravenous infusions dosed at 0.5mg/kg.
Behavioral: Minimally Enhanced Usual Care — Minimally Enhanced Usual Care will consist of educational reading materials regarding chronic back pain and depression and will be provided to participants in arms 2 and 3 (pilot RCT).
  Other Names: Control
  Arms: Intervention + Minimally Enhanced Usual Care; Minimally Enhanced Usual Care Only
Behavioral: Brief narrative intervention — Participants in Arm 1 (open label pilot) will receive the brief narrative intervention after four ketamine infusions.
  Participants in Arm 2 (those randomized after ketamine infusions are complete to the active arm of the pilot RCT) will receive the brief narrative intervention.
  Other Names: Active/intervention
  Arms: Intervention + Minimally Enhanced Usual Care; Open label, single arm pilot

SUMMARY:
This is a pilot study to evaluate the feasibility, acceptability, and safety of ketamine infusions followed by a brief behavioral intervention in Veterans with chronic low back pain and depression.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) and depression are top causes of disability in the United States. Veterans are more likely to have both; prevalence is increasing. When CLBP and depression occur together, patients report more functional limitations, unemployment, and higher healthcare spending, and treatment is less successful. Novel approaches simultaneously addressing pain interference and depression symptoms are needed.

This study will involve initial pilot feasibility testing of an intervention designed to help participants with chronic low back pain and depression both reduce pain interference and improve mood. This study will occur in two phases. The initial phase is a open-label single-arm pilot of the combined intervention (ketamine infusions followed by the brief behavioral intervention) in a small sample of Veterans (n=5). The objective is to develop and assess initial feasibility of study procedures and obtain participant feedback through semi-structured exit interviews. The second phase consists of a single-blind, two-arm, pilot feasibility randomized controlled trial (RCT) (n=44, 22 per arm) which will (a) assess feasibility benchmarks and (b) collect outcome data that will be used to calculate sample size to power a larger RCT.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with self-report of moderate to severe, high impact chronic low back pain (defined as 4/10 in severity via NRS, present 3 months on most days) and associated pain interference (defined as T-score 60 on the PROMIS Pain Interference measure), and current significant depressive symptoms (defined as a score 11 on the Quick Inventory of Depressive Symptoms - Self Report (QIDS-SR).
* Medically stable (no hospitalizations in the past month lasting 3 days).
* No changes in pain or depression medication regimen in 4 weeks.
* No planned surgery, injections, hospitalizations, or other new interventions for back pain (except for physical therapy or exercise) or depression during the next four months (study duration).
* Participants must have an adult who can drive them home after the ketamine treatments.

Exclusion Criteria:

* Inability to speak English due to the narrative intervention being conducted in English.
* Inability or unwillingness to provide written informed consent (e.g. current delirium).
* Current psychotic symptoms, or history of schizophrenia, schizoaffective disorder, and other psychotic disorder.
* Currently participating in another clinical trial for pain or depression.
* Current uncontrolled hypertension (defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg).
* Known elevated intracranial pressure, cerebral arterial aneurysm, or elevated intraocular pressure.
* History of cirrhosis or unstable cardiac condition (e.g., decompensated congestive heart failure).
* Any of the following lab values >2x upper limit of normal: alanine transaminase (ALT), aspartate transferase (AST), direct bilirubin, alkaline phosphatase, creatinine; thyroid stimulating hormone (TSH) <2x lower limit of normal or >2x upper limit of normal.
* Positive urine pregnancy test or lack of birth control method in Veterans of childbearing potential.
* Known hypersensitivity to any excipient in the ketamine injection formulation.
* Previously experienced serious adverse effects with ketamine.
* On day of ketamine infusions, a urine drug screen positive for non-prescribed substances(s) (except cannabis) will exclude a participant from receiving ketamine
* Current or previous abuse of ketamine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Interference (PROMIS Short Form v1.1 Pain Interference 6b) | Visit 7 (8-10 days post randomization)
  Pain interference, defined as the extent to which pain impedes enjoyment of and participation in life activities (including cognitive, social, recreational, and self-care activities), will be the primary outcome. Raw scores (range 6 - 30, higher scores indicating more interference) are normed to mean of general population (T-score 50; SD 10); higher T-scores indicate higher pain interference. Minimum clinically important change is 3.0 - 3.5 point reduction in the T-score.

SECONDARY OUTCOMES:
Pain intensity (Numeric Rating Scale) | Visit 7 (8-10 days post randomization)
  Pain intensity will be measured using the NRS, a single-item measure where participants rate their pain intensity on a scale of 0 (no pain) to 10 (worst pain imaginable). In chronic pain, a reduction of 2 points or 30% is considered a meaningful improvement.
Depression (Quick Inventory of Depressive Symptoms - Self Report (QIDS-SR) ) | Visit 7 (8-10 days post randomization)
  The Quick Inventory of Depressive Symptoms - Self Report (QIDS-SR) is a 16-item rating scale assessing self-report of depressive symptoms. Scores range from 0 - 27, with higher scores indicating more severe depressive symptoms. Reductions of approximately 30% are considered clinically meaningful improvements in depressive symptoms.

OTHER OUTCOMES:
Feasibility - Enrollment | 18 months from start of study
  Enrollment benchmarks involve aiming to enroll 2-4 participants/month.
Presence of adverse events (AE)s | Visits 1-7 or weekly (whichever is more frequent); Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Safety will be assessed via Adverse event (AE) assessment which will be obtained by means of a standard form assessing the presence of AEs.
Pain Interference (PROMIS Short Form v1.1 Pain Interference 6b) | Visit 1 (Baseline), Visit 5 (post ketamine pre randomization), Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Pain interference will also be measured at these additional time points. Participants rate each item regarding experiences over the past 7 days on a Likert scale from 1 (not at all) to 5 (Very much). Raw scores (range 6 - 30, higher scores indicating more interference) are normed to mean of general population (T-score 50; SD 10); higher T-scores indicate higher pain interference. Minimum clinically important change is 3.0 - 3.5 point reduction in the T-score.
Pain Intensity (Numeric Rating Scale) | Visit 1 (Baseline), Visit 5 (post ketamine pre randomization), Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Pain intensity will also be measured at these additional time points. Pain intensity will be measured using the NRS, a single-item measure where participants rate their pain intensity on a scale of 0 (no pain) to 10 (worst pain imaginable). In chronic pain, a reduction of 2 points or 30% is considered a meaningful improvement.
Depression (Quick Inventory of Depressive Symptoms - Self Report (QIDS-SR) ) | Visit 1 (Baseline), Visit 5 (post ketamine pre randomization), Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Depression will also be measured at these additional time points.
Acceptability | Visit 7 (8-10 days post randomization)
  Participants will rate acceptability in multiple domains (helpfulness; convenience and comfort; satisfaction) on a 1-4 scale (1=very dissatisfied, 2=somewhat dissatisfied, 3=somewhat satisfied, 4=very satisfied). Benchmarks for acceptability include >70% "somewhat" or "very satisfied" in all domains.
Global Impression of Change (Patient Global Impression of Change (PGIC)) | Visit 7 (8-10 days post randomization), Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Participants rate their change overall on a 7-point Likert scale ranging from 1 (very much improved) to 7 (very much worse).
Cognitive Flexibility (Cognitive Flexibility Scale (CFS)) | Visit 1 (Baseline) , Visit 5 (post ketamine infusions pre randomization), Visit 7 (8-10 days post randomization), Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Cognitive flexibility refers to individuals' awareness of alternatives to a given situation, willingness to consider them, and belief that they can adapt. Individuals rate 12-items of the Cognitive Flexibility Scale (CFS) on a 6 point Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree), total score range 12 - 72. Higher scores indicate more cognitive flexibility.
Psychological Flexibility (Emotion Regulation Questionnaire (ERQ-9)) | Visit 1 (Baseline) , Visit 5 (post ketamine infusions pre randomization), Visit 7 (8-10 days post randomization), Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Psychological flexibility refers to individuals' ability to both recognize and accept emotions and choose their subsequent action based on core beliefs and values (rather than a reflexive emotional response). It will be assessed via the 9-item Emotion Regulation Questionnaire (ERQ-9).
Psychological Inflexibility (Acceptance and Action Questionnaire-II (AAQII)) | Visit 1 (Baseline) , Visit 5 (post ketamine infusions pre randomization), Visit 7 (8-10 days post randomization), Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Psychological inflexibility will be assessed by the 7-item Acceptance and Action Questionnaire-II (AAQII).
Psychologically insightful experiences occurring in response to ketamine administration (Psychological Insight Questionnaire (PIQ)) | Visit 5 (post ketamine infusions pre randomization)
  The Psychological Insight Questionnaire (PIQ) is a 23-item questionnaire developed to assess acute discoveries or realizations occasioned by a psychedelic experience, such as those regarding one's personality, relationships, behavioral patterns, or emotions. We will use the PIQ to assess changes in response to ketamine.
Mystical Experiences Occasioned by Ketamine (Mystical Experience Questionnaire (MEQ)) | Visit 5 (post ketamine infusions pre randomization)
  The Mystical Experience Questionnaire (MEQ) is a 30-item validated measure assessing 4 factors of a mystical or psychedelic experience occasioned by ketamine. These include a mystical experience (e.g., "freedom from the limitations of your personal self and feeling a unity or bond with what was felt to be greater than your personal self"), positive mood (e.g., "sense of awe or awesomeness"), transcendence of time and space, and ineffability (feeling that the experience cannot be conveyed in words).
Catastrophizing (Catastrophizing Subscale from the Coping Strategies Questionnaire (CSQ-CAT)) | Visit 1 (Baseline) , Visit 5 (post ketamine infusions pre randomization), Visit 7 (8-10 days post randomization), Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Catastrophizing (the tendency to think of the future as irrationally negative) associates with poor outcomes in the setting of chronic pain, including poorer functional status. It will be measured via the 6-item Catastrophizing Subscale from the Coping Strategies Questionnaire (CSQ-CAT).
Self-Efficacy (PROMIS Self-Efficacy for Chronic Conditions - Managing Daily Activities -Short Form 4a) | Visit 1 (Baseline) , Visit 5 (post ketamine infusions pre randomization), Visit 7 (8-10 days post randomization), Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Self-efficacy is a cognitive tendency to perceive oneself as capable of managing life's problems. It will be measured via the 4-item PROMIS Self-Efficacy for Chronic Conditions - Managing Daily Activities -Short Form 4a.
Fear-Avoidance Beliefs/Kinesiophobia (Fear-Avoidance Beliefs Questionnaire-Physical Activity Subscale (FABQ-PA)) | Visit 1 (Baseline) , Visit 5 (post ketamine infusions pre randomization), Visit 7 (8-10 days post randomization), Visit 8 (1 month follow up), Visit 9 (3 month follow up)
  Fear-avoidance beliefs refers to the cognitive appraisal that certain kinds of activities may cause additional damage or pain; more fear-avoidance beliefs for physical activity (also called kinesiophobia) predict development of chronic pain and disability in those with acute low back pain. Fear-avoidance beliefs will be measured using the 4-item Fear-Avoidance Beliefs Questionnaire-Physical Activity Subscale (FABQ-PA).
Nociplastic Pain Characteristics (Fibromyalgia Survey Questionnaire (FSQ)) | Visit 1 (Baseline)
  The Fibromyalgia Survey Questionnaire (FSQ), adapted from the American College of Rheumatology Fibromyalgia Survey score, will be used to measure pain widespreadness and accompanying symptoms, also known as nociplastic features. It consists of two scales, the Widespread Pain Index (WPI) and the Symptom Severity score (SSS). The WPI instructs participants to indicate location(s) of pain (range 0 - 19, higher scores indicate more areas of pain). The SS score assesses additional symptoms including fatigue, unrefreshing sleep, and cognitive disruption (range 0 -12, higher scores indicate more symptoms). Total score range is 0 - 31, with higher scores indicating more nociplastic features of pain. Fibromyalgia screening positive cut points are WPI >=7 and SSS >=5 OR WPI of 4-6 and SSS >= 9.
Neuropathic Pain Characteristics (painDETECT) | Visit 1 (Baseline)
  PainDETECT will be used to evaluate presence of neuropathic features of back pain. PainDETECT instructs individuals to rate pain at different time points (range 0 - 10, with higher scores indicating more severe pain), and to select/rate agreement with items on a Likert scale from never to very strongly. Total score range is 0 - 38, with those scoring >18 having likely neuropathic components of back pain.
Feasibility - retention/attendance | Visit 7 (8-10 days post randomization)
  Target >70% of participants who complete baseline measures will complete all four ketamine infusion sessions, the behavioral intervention (if assigned) and the initial post-intervention assessment battery.
Feasibility - measurement completion | Visit 9 (3 month follow up)
  Target >80% of participants complete follow-up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria D Powell, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No